CLINICAL TRIAL: NCT03989388
Title: Occupational Self-Analysis Programme in Participants With Intellectual Disabilities, Acquired Brain Injury and Students
Brief Title: Occupational Self-Analysis Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, María Rodríguez Bailón, Principal investigator, University of Malaga
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Occupational Self-Analysis2016
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Occupational Therapy; Intellectual Disability; Acquired Brain Injury; Students; Stroke; Awareness
MeSH Terms: conditions — Intellectual Disability; Brain Injuries; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Occupational Self-Analysis Programme
  Interventions: Behavioral: Occupational self-analysis
- Control group (Active Comparator): Vocational guidance or usual rehabilitation (in the case of ABI participants)
  Interventions: Behavioral: Vocational guidance; Behavioral: Usual Rehabilitation

INTERVENTIONS:
Behavioral: Occupational self-analysis — The "Occupational Self-Analysis" program provides participants with a space where they can learn to analyse the barriers and supports for occupational participation.
  Arms: Intervention Group
Behavioral: Vocational guidance — To explore participant´s job interests and learned how to find a job and define a professional profile.
  Arms: Control group
Behavioral: Usual Rehabilitation — Usual rehabilitation: occupational therapy and/or physiotherapy.
  Arms: Control group

SUMMARY:
Introduction There is a growing tendency from Occupational Therapy towards the use of programs based on occupation, which, through significant occupational participation, have shown to obtain beneficial results maintained over time in its participants. For this, these programs carry out processes of occupational self- analysis in which people reflect on the daily activities they usually perform so that they can generate modifications towards more satisfactory routines. However, and despite their proven benefits, these programs have been conducted mainly on older people and in cultural contexts other than Spanish.

The "Occupational Self-Analysis" program, developed in the Spanish context, provides participants with a space where they can learn to analyse the barriers and supports for occupational participation and thus achieve a more significant occupational performance.

Objectives The objective of this study was to assess the effectiveness of the "Occupational Self-Analysis" program on the subjective perception of health and the number of roles in people with and without disabilities. In the same way, the purpose was to analyse the increase or modification of the performance in the Activities of the Daily Life that the participants did, and to know how the social environment supports the individual participation of the participants in meaningful activities.

Method The implementation of the "Occupational Self-Analysis" program was carried out in 3 different populations; people with intellectual disability, people with acquired brain injury (ABI) and University students. The intervention was performed by comparing it with a control group (vocational guidance or usual rehabilitation in the caso of ABI participants). In people with intellectual disability, the experimental group consisted of 12 participants and the control one of 13. In people with ABI, the experimental group involved 5 participants and the control, 7. In university students, the experimental group involved 7 and the control 7. The SF-36 Health Questionnaire was used for the evaluation of subjective health perception and the Roles Checklist (Part 1) to evaluate the number of roles they play in the present and the future. All of them underwent a final focus group and the diary were they wrote their learning and emotions was analyzed to assess the benefits of the program.

DETAILED DESCRIPTION:
Results A positive trend was observed in all dimensions of the SF-36 Health Questionnaire in people with intellectual disability and ABI. In the experimental group of people with intellectual disability the improvements were significant compared to the control group in the dimensions of role limitations due to physical problems (Z = -2.41, p = .016), role limitations due to emotional problems (Z = - 1.99; p = .046), social function (Z = -3.35; p = .001) and the accumulated scores of the mental component (Z = -2.66; p = .008). On the other hand, the ABI experimental group obtained significant improvements in vitality after the intervention (Z = -2.20, p = .028), not finding statistically significant improvements compared to the control group.

With respect to the number of roles internalized, both the experimental group with intellectual disability and the one presenting ABI experienced a marginally significant increase in the number of roles that participants wanted to develop in the future after taking part in the program.

Both in people with intellectual disability, ABI and students, the program improved the involvement in meaningful activities through the inclusion of new occupations, modification of previous habits or the transformation of solitary activities into social participation activities. In addition, the participants increased their awareness of those factors that influenced their participation in meaningful activities. This meant becoming aware of aspects related to volition, habituation, personal abilities and the environment.

ELIGIBILITY:
Participants with Intellectual disabilities:

Inclusion Criteria:

- Basic skills such as writing, reading or calculation

Exclusion Criteria:

-Unsuitable social behaviour

Participants with Acquired Brain Injury:

Inclusion Criteria:

- Members of an association for people with neurological impairment.

Exclusion Criteria:

* Behavioral problems
* Problems speaking or understanding.

Students:

Inclusion Criteria:

- Occupational therapy student.

Exclusion Criteria:

* Absenteeism
* Lack of suitable social behavior

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
SF-36 Health Questionnaire | 30 minutes
  Evaluation of subjective health perception.
  Variables:
  * Eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
  * Physical component summary (Mean scores of four domains: physical functioning, role limitations caused by physical health problems, bodily pain, and general health) (Range 0-100)
  * Mental component summary scores (Mean scores of four domains: role limitations caused by emotional problems, vitality, social functioning, and mental health) (Range 0-100)
Roles Checklist | 20 minutes
  Past, present and future occupational roles (Part 1 of Roles Checklist). Variables:
  - Number of roles in each period (Range 0-10).
Focus groups | 1 hour
  Qualitative data: Perceived learning and emotions
Participant diary | 2 hours
  Perceived learning and emotions in a participant diary after sessions

CONTACTS AND LOCATIONS:
Overall Officials: Ana Judit Fernández-Solano, PhD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (2):
- Spain (2):
  - Asociación de Daño Cerebral de Málaga (ADACEMA), Málaga
  - Universidad Católica San Antonio de Murcia, Murcia

REFERENCES:
- [Background] Fernandez-Solano AJ, Del Bano-Aledo ME, Rodriguez-Bailon M. From thinking to acting: occupational self-analysis tools for use with people with intellectual disability. A pilot study. J Intellect Disabil Res. 2019 Sep;63(9):1086-1096. doi: 10.1111/jir.12621. Epub 2019 Apr 24. PMID 31017354